CLINICAL TRIAL: NCT01832246
Title: Prospective Study of Endoscopic Ultrasonographic Staging and Conventional Endoscopic Staging for Depth of Invasion and Endoscopic Tumor Size Estimation for Early Gastric Cancer
Brief Title: Endoscopic Ultrasonographic Staging and Conventional Endoscopic Staging for Depth of Invasion for Early Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeongmin Choi, professor, Department of Internal Medicine and Liver Research Institute, Seoul National University Hospital
Other Study IDs: 20122012
Record Dates: First submitted 2012-07-04; First posted 2013-04-16 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Gastric Tumor; Early Gastric Cancer
Keywords: endoscopy; endosonography; stomach cancer; tumor staging
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The accurate prediction of depth of tumor invasion in early gastric cancer is essential for the proper selection of candidates for endoscopic resection. Conventional endoscopy and endoscopic ultrasonography have been useful diagnostic method for depth of invasion in early gastric cancer. However, there has been no prospective comparative study on the accuracy between the 2 methods. Therefore, the investigators prospectively compare the accuracy between the 2 methods regarding prediction of depth of invasion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with early gastric adenocarcinoma undergo both endoscopic staging and endoscopic ultrasonographic staging for depth of invasion

Exclusion Criteria:

* patients had previously received neoadjuvant chemotherapy or chemoradiotherapy
* patients with obviously advanced gastric cancer by endoscopy
* the evidence of distant metastasis or extensive adjacent organ invasion on abdominal CT scan

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with early gastric adenocarcinoma is prospectively enrolled at Seoul National University Hospital.
Sampling Method: Probability Sample
Enrollment: 560 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy between endoscopic ultrasonographic staging and conventional endoscopic staging | up to 2.5 years (end of study, December 2014)

CONTACTS AND LOCATIONS:
Overall Officials: Sang Gyun Kim, M.D., Study Director — Department of Internal Medicine and Liver Research Institute, Seoul National University College of Medicine; Jeongmin Choi, M.D., Principal Investigator — Department of Internal Medicine and Liver Research Institute, Seoul National University College of Medicine
Locations (1):
- Division of Gastroenterology, Department of Internal Medicine and Liver Research Institute, Seoul National University Hospital, Seoul, Seoul, South Korea